CLINICAL TRIAL: NCT06383429
Title: Relation Between Forward Head Posture and Incidence of Headache in Obese Adults
Status: Completed | Type: Observational
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Ababa, lecturer of internal physical therapy, Ahram Canadian University
Other Study IDs: P.T-WH-10/2023-521
Record Dates: First submitted 2024-04-21; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Obese; Headache; Neck Pain
MeSH Terms: conditions — Obesity; Headache; Neck Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: forward head posture by using mobile application. And patients will fill out headache disability index. — forward head posture by using mobile application. And patients will fill out headache disability index.

SUMMARY:
Cross sectional study to detect relation between forward head posture and headache. We will take information from the patient about:

* Detailed history of patient
* Forward head posture by using mobile application
* Headache disability index

ELIGIBILITY:
Inclusion Criteria:

* obese adult with forward head posture

Exclusion Criteria:

* any neurological condition , autoimmune diseases and cervical disc

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: obese adulty with forward head posture
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
forward head posture | one time
  mobile application asses forward head posture
BMI | one time
  body mass index to detect obesity
headache disability index | one time
  to asses seversity of headache

CONTACTS AND LOCATIONS:
Locations (1):
- Ababa physical therapy center, Banī Suwayf, Beni- Suaf, Egypt

IPD SHARING:
Plan to Share IPD: No